CLINICAL TRIAL: NCT02835833
Title: Phase I Dose Escalation Study of Nintedanib Plus Bevacizumab in Advanced Solid Tumors
Brief Title: Study of Nintedanib Plus Bevacizumab in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Francisco Robert,MD, Professor, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F160202011 (UAB 15108)
Record Dates: First submitted 2016-07-07; First posted 2016-07-18 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Renal Cell Carcinoma; Colorectal Adenocarcinoma; Non-squamous Non-small Cell Lung Cancer; Platinum-refractory Ovarian Carcinoma; Cervical Carcinoma
Keywords: advanced solid tumors; Nintedanib; Bevacizumab; dose escalation
MeSH Terms: conditions — Carcinoma, Renal Cell; Uterine Cervical Neoplasms | interventions — nintedanib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nintedanib 150 mg + Bevacizumab 15 mg/kg (Experimental): The first three patients on study will be treated with 150 mg orally of Nintedanib two times daily plus 15 mg/kg of Bevacizumab administered intravenously on day one of each three week cycle.
  If one dose limiting toxicity occurs in the first cohort, then three more patients will be treated at that same starting dose and assessed for toxicity after cycle two. If two or more patients have dose limiting toxicity, then dose escalation will end and the maximum tolerated dose will be reached.
  Interventions: Drug: Nintedanib; Drug: Bevacizumab
- Nintedanib 200 mg + Bevacizumab 15 mg/kg (Experimental): If no patients experience dose limiting toxicity, then three additional patients will be treated with 200 mg orally of Nintedanib two times daily plus 15 mg/kg of Bevacizumab administered intravenously on day one of each three week cycle.
  Interventions: Drug: Nintedanib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Nintedanib — Nintedanib will be given twice daily at either 150 mg or 200 mg.
  Other Names: BIBF1120
Drug: Bevacizumab — Bevacizumab will be given at 15 mg/kg
  Other Names: Avastin

SUMMARY:
Angiogenesis, the development of new blood vessels, plays an important role in the disease development and tumor growth in many solid organ malignancies. Bevacizumab was the first anti-angiogenic drug to be approved in solid tumors and has shown advantageous activity with multiple tumor types. However, the responses from Bevacizumab are often transient due to the tumor's manipulative abilities to circumvent the usual pathways to find salvage pathways instead.

Nintedanib has demonstrated anti-tumor activity in non-squamous non-small cell lung cancer, colorectal cancer, ovarian cancer, and renal cell cancer. The combination of Bevacizumab and Nintedanib are being proposed to target the tumor's manipulation processes to generate alternate pathways for angiogenesis thus creating a potential benefit to delay tumor growth.

DETAILED DESCRIPTION:
This is an open-label, phase I dose-escalation study of Nintedanib combined with standard-dose Bevacizumab for advanced solid tumors in which Bevacizumab has an indication. The primary endpoints will be safety and tolerability of the drug combination and a determination of recommended Phase II dose for Nintedanib in combination with standard dose Bevacizumab.

The first three patients will be treated with Nintedanib daily plus Bevacizumab on day one of each three week cycle. If there are no dose limiting toxicities, then three additional patients will be treated with the same drugs with Nintedanib at a slightly higher level. Finally, a third cohort of three patients will be dosed at an even higher level. Once the maximum tolerated dose of Nintedanib is reached, then an additional six patients will be treated at that dose in combination with Bevacizumab until disease progression or unacceptable toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Histologically proven advanced or metastatic solid cancer for which Bevacizumab has an indication: renal cell carcinoma, colorectal adenocarcinoma, non-squamous non-small cell lung cancer, platinum- refractory ovarian carcinoma, cervical carcinoma.
3. Life expectancy at least 3 months
4. ECOG performance status score 0-1
5. Progression after at least first-line systemic therapy for metastatic disease
6. At least one measurable lesion according to RECIST criteria or any other baseline prerequisite for the assessment of the principal judgement criteria.
7. Signed and dated written informed consent prior to admission to the study
8. Resolution of all acute adverse events resulting from prior cancer therapies to NCI CTCAE grade less than/equal to 1 or baseline (except alopecia)
9. Adequate organ function as defined by the following criteria

   * AST/ALT ≤ 2.5x upper limit of normal (ULN) in the case of liver metastases or AST/ALT ≤ 1.5 x ULN in patients without liver metastases
   * total serum bilirubin within normal limits regardless of liver metastases
   * absolute neutrophil count (ANC) > 1500
   * Platelets > 100k without transfusion support in the past 28 days
   * Hemoglobin > 9.0 without transfusion support in the past 28 days
   * Serum creatinine < 1.5x ULN
   * Prothrombin time/INR and partial thromboplastin time within normal limits
   * Urinalysis ≤ 1+ protein
10. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

1. Previous therapy with Bevacizumab is allowed, but patient who experienced serious dose-limiting toxicities while on prior Bevacizumab therapy are excluded
2. Prior treatment with Nintedanib (BIBF1120). Known hypersensitivity to Nintedanib, peanut or soya or any other trial drug, their excipients or to contrast media
3. Chemo-, hormone-, radio-(except for brain and extremities) or immunotherapy or therapy with monoclonal antibodies or small tyrosine kinase inhibitors within the past 4 weeks prior to treatment with the trial drug.
4. Radiotherapy to the target lesion within the past 3 months prior to baseline imaging
5. Persistence of clinically relevant therapy related toxicity from previous chemo and/or radiotherapy
6. History of brain involvement with cancer, spinal cord compression, carcinomatous meningitis, or new evidence of brain or leptomeningeal disease. Patients with irradiated or resected brain lesions are permitted provided the lesions are fully treated and inactive, patients are asymptomatic, and no steroids have been used for at least 28 days.
7. Leptomeningeal disease
8. Centrally located tumours with radiographic evidence of local invasion of major blood vessels
9. Treatment with other investigational drugs or treatment in another clinical trial within the past 4 weeks before start of therapy or concomitantly with the trial
10. Therapeutic anticoagulation (except low-dose heparin and/or heparin flush as needed for maintenance of an in-dwelling intravenous devise) or anti-platelet therapy (except for low-dose therapy with acetylsalicylic acid <325mg per day.
11. Major injuries and/or surgery within the past 4 weeks prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period.
12. History of clinically significant hemorrhagic or thromboembolic event in the past 6 months.
13. Known inherited predisposition to bleeding or thrombosis
14. Significant cardiovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within the past 6 months prior to start of study treatment, congestive heart failure >New York Heart Association II, serious cardiac arrhythmia, pericardial effusion)
15. Proteinuria CTCAE grade 2 or greater
16. Creatinine >1.5 ULN or GFR <45 ml/min
17. Hepatic function: total bilirubin outside of normal limits; ALT or AST >2.5 ULN in pts without liver metastasis. For patients with liver metastasis: total bilirubin outside of normal limits, ALT or AST >5 x ULN
18. Coagulation parameters: International normalized ratio (INR) >2, prothrombin time (PT) and partial thromboplastin time (PTT) >50% of deviation of institutional ULN
19. Absolute neutrophil count (ANC) <1500/ml, platelets <100,000/ml, Hemoglobin <9.0 g/dl
20. Other malignancies within the past 5 years other than basal cell skin cancer or carcinoma in situ of the cervix
21. Active serious infections in particular if requiring systemic antibiotic or antimicrobial therapy
22. Active or chronic hepatitis C and/or B infection
23. Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
24. Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study.
25. Patients who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) during the trial and for at least three months after end of active therapy.
26. Pregnancy or breast feeding. Female patients must have a negative pregnancy test (β-HCG test in urine or serum) prior to commencing study treatment and must agree with the use of effective contraception during the study and for three months following last dose of Nintedanib.
27. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule
28. Active alcohol or drug abuse
29. Minor surgical procedures such as Mediport placement or core biopsies within 7 days of study treatment
30. Stroke, transient ischemic attack, arterial embolism, percutaneous transluminal coronary angioplasty (PTCA), or coronary artery bypass grafting (CABG) within the past 6 months
31. History of pulmonary hemorrhage or hemoptysis within 6 months of starting study treatment
32. Open wounds or unhealed fractures within 28 days of starting study treatment
33. Known HIV or AIDS related illness

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-06-09 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2018-06-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Initial dose of study drug until four weeks after the last dose or until death, whichever occurs first
  Adverse event reporting will be graded following the National Cancer Institute of Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.
Maximum tolerable dose of Nintedanib | Baseline up to three years
  The maximum dosage of drug that yields acceptable toxicity levels.

SECONDARY OUTCOMES:
Objective tumor response rate | up to 100 weeks
  Response will be evaluated using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
Progression-free survival | Baseline up to three years
  Progression-free survival is defined as the duration of time from start of treatment to the first documentation of tumor progression. Kaplan-Meier estimates will be used.
Plasma level of vascular endothelial growth factor (VEGF) | Baseline up to two years
  Correlative analysis will be conducted using Chi-square tests and Spearman rank correlations. Differences between responders and non-responders will utilize the Kruskal-Wallis test.
Plasma level of platelet-derived growth factor (PDGF) | Baseline up to two years
  Correlative analysis will be conducted using Chi-square tests and Spearman rank correlations. Differences between responders and non-responders will utilize the Kruskal-Wallis test.
Plasma level of vascular endothelial growth factor and receptor (VEGF-R) | Baseline up to two years
  Correlative analysis will be conducted using Chi-square tests and Spearman rank correlations. Differences between responders and non-responders will utilize the Kruskal-Wallis test.
Plasma level of phosphatidylinositol-glycan biosynthesis class F protein (PIGF) | Baseline up to two years
  Correlative analysis will be conducted using Chi-square tests and Spearman rank correlations. Differences between responders and non-responders will utilize the Kruskal-Wallis test.
Plasma level of fibroblast growth factor (FGF) | Baseline up to two years
  Correlative analysis will be conducted using Chi-square tests and Spearman rank correlations. Differences between responders and non-responders will utilize the Kruskal-Wallis test.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Robert, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paluri R, Madan A, Li P, Jones B, Saleh M, Jerome M, Miley D, Keef J, Robert F. Phase 1b trial of nintedanib in combination with bevacizumab in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2019 Mar;83(3):551-559. doi: 10.1007/s00280-018-3761-y. Epub 2019 Jan 2. PMID 30603797